CLINICAL TRIAL: NCT00561262
Title: An Evaluation of Hemi-ablation Therapy Using High-Intensity Focused Ultrasound in the Treatment of Localized Adenocarcinoma of the Prostate
Brief Title: High-Intensity Focused Ultrasound Therapy in Treating Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000574367; UCLCTC-UCLH-HEMI-HIFU; EU-20774; ISRCTN25145525
Record Dates: First submitted 2007-11-17; First posted 2007-11-20 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Intensity Focused Ultrasound Ablation

INTERVENTIONS:
Other: questionnaire administration
Procedure: high-intensity focused ultrasound ablation
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: High-intensity focused ultrasound energy may be able to kill tumor cells by heating them without affecting normal tissue.

PURPOSE: This phase II trial is studying how well high-intensity focused ultrasound ablation therapy works in treating patients with localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine patient acceptability, feasibility, and side-effect profile by evaluating records of adverse events.
* To determine patient acceptability, feasibility, and side-effect profile by evaluating urinary symptoms and erectile function before study stage 1 (verification), before study stage 2 (treatment), and at each follow-up visit.

Secondary

* To determine the effectiveness of therapy by post-treatment transrectal ultrasound-guided biopsies at 6 months and if there is evidence of biochemical failure.
* To determine the effectiveness of therapy by post-treatment MRI to evaluate area of necrosis and presence of any residual tissue.
* To determine the effectiveness of therapy by measurement of prostate-specific antigen (PSA) at each follow-up visit and measurement of time to PSA nadir.
* To determine the effectiveness of therapy by recording the need for secondary or adjuvant treatment following therapy.

OUTLINE: Patients undergo hemiablation using high-intensity focused ultrasound to the side of the prostate with cancer and up to 5 mm over into the contralateral side to ensure adequacy.

Patients complete questionnaires periodically during study to assess urinary symptoms and erectile dysfunction. These include the International Index of Erectile Function-15 [IIEF-15]; the International Prostate Symptom Score [IPSS] and IPSS-QoL; the Functional Assessment of Cancer Therapy - Prostate (FACT-P); and the Continence Questionnaire.

After completion of study treatment, patients are followed at 2-7 days, 7-14 days, and at 1, 3, 6, 9, and 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate, meeting the following criteria:

  * Gleason score ≤ 7 (patterns 3+4 or 4+3 or less are acceptable)
  * Cancer prostate-confined only
  * Cancer confined to one lobe as defined by transrectal ultrasound (TRUS) biopsy
  * Serum prostate-specific antigen (PSA) ≤ 15 ng/mL
  * Prostate volume ≤ 40 cc OR AP length of prostate < 4 cm
* Unilateral prostate adenocarcinoma must be verified in stage 1 of this trial unless the patient has had multi-sequence MRI and transperineal template biopsies outside of this trial in similar procedure protocols to this trial
* No evidence of metastatic disease
* No intraprostatic calcifications ≥ 10 mm in size in cancer-positive side of prostate

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 5 years
* No latex allergies
* No American Society of Anesthesiology surgical risk score III or IV
* No contraindications to MRI scanning (e.g., severe claustrophobia, permanent cardiac pacemaker, or metallic implant likely to contribute significant artefact to images)
* Must be fit for general anesthesia or regional anesthesia as assessed by the consultant anesthetist

PRIOR CONCURRENT THERAPY:

* More than 6 months since prior androgen suppression therapy
* No prior radiotherapy for prostate cancer
* No prior chemotherapy for prostate cancer
* No prior significant rectal surgery preventing insertion of transrectal probe
* No prior transurethral resection of the prostate or laser prostatectomy
* No prior high-intensity focused ultrasound, cryosurgery, thermal, or microwave therapy to the prostate

Max Age: 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-10 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Feasibility
Adverse events
Patient acceptability as assessed by Assessment of Cancer Therapy - Prostate (FACT-P), International Prostate Symptom Score (IPSS) , IPSS-Quality of Life, Continence Questionnaire, and 15-Item International Index of Erectile Function
Side effect profile

SECONDARY OUTCOMES:
Measurement of prostate-specific antigen (PSA) kinetics including time to PSA nadir
Exclusion of cancer on MRI at 2-7 days and at 6 months
Transrectal ultrasound biopsies at 6 months
Need for secondary or adjuvant treatment for prostate cancer following therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mark Emberton, MD, FRCS, MBBS, Study Chair — University College London Hospitals
Locations (1):
- University College of London Hospitals, London, England, United Kingdom

REFERENCES:
- [Result] Ahmed HU, Freeman A, Kirkham A, Sahu M, Scott R, Allen C, Van der Meulen J, Emberton M. Focal therapy for localized prostate cancer: a phase I/II trial. J Urol. 2011 Apr;185(4):1246-54. doi: 10.1016/j.juro.2010.11.079. Epub 2011 Feb 22. PMID 21334018